CLINICAL TRIAL: NCT01349920
Title: An Open Label Study to Discover Biomarkers of Intestinal Mucosal Healing in Crohn's Disease (CD)
Brief Title: Biomarkers of Intestinal Mucosal Healing in Crohn's Disease (P08143)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P08143; 2011-000517-40 (EudraCT Number); MK-2155-195
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Crohn Disease
Keywords: biological markers; endoscopy; gastrointestinal
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool, serum, peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab 5 mg/kg: Infliximab treatment and endoscopy.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab administered intravenously at a dose of 5 mg/kg at study Weeks 0, 2, 6, 14, and 22.
  Other Names: Remicade; SCH 215596; MK-2155

SUMMARY:
This study will evaluate biomarkers that reflect changes in gut mucosal status during therapy with infliximab and determine whether changes in the levels of the selected biomarkers can be used to predict endoscopically assessed gut mucosal status changes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohn's Disease (CD) of at least 6 weeks duration, or acute diagnosis of sufficiently severe CD warranting initiation of infliximab sooner than allowed by fecal calprotectin turnaround time
* History of colonic involvement verified by prior endoscopy or radiography
* Indicated for treatment with infliximab according to current best medical practice
* Body Mass Index (BMI) between 15 kg/m^2 and 35 kg/m^2
* Women of childbearing potential and non-vasectomized men agree to use medically-acceptable contraception
* Negative pregnancy test
* No signs or symptoms of active tuberculosis (TB) and has a negative TB test within 6 weeks of first study drug administration

Exclusion Criteria:

* Pregnancy, intention to become pregnant, or breastfeeding
* Evidence of a colon unaffected by CD
* Indication for surgery
* Perianal disease likely to interfere with study participation
* Presence of a stoma or history of colectomy
* Symptomatic diarrhea unrelated to CD
* Strictures or evidence of bowel obstruction
* Presence of abscess unless completed definitive treatment can be documented one week prior to screening
* Presence of fistulas
* Contraindication to infliximab
* Intolerance to sedatives or other medications required for endoscopy
* Any prior use of anti-inflammatory biologic therapy
* Moderate or severe congestive heart failure
* History of demyelinating disease or symptoms suggestive of multiple sclerosis or optic neuritis
* Major surgery or donation/loss of at least one unit of blood within 4 weeks of screening
* Positive for hepatitis B surface antigen, hepatitis C antibodies, or Human Immunodeficiency Virus (HIV)
* History of any tumor except adequately treated basal cell carcinoma or carcinoma in situ of the cervix
* History of systemic granulomatous infection
* History of nontuberculous mycobacterial disease, or any opportunistic infection within 12 months of study entry
* Transplanted organ including bone marrow or hematopoietic stem cell-derived marrow

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Approximately 20 participants aged 18 to 60 years with Crohn's Disease will be enrolled from gastrointestinal specialist clinics.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2015-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants 18 to 60 years of age, with moderate to severe Crohn's Disease (CD) who had not been previously treated with anti-inflammatory biologic agents were enrolled in this trial.
Groups:
- Infliximab 5mg/kg: Infliximab administered intravenously at a dose of 5 mg/kg at study weeks 0, 2, 6, 14, and 22
Period: Overall Study
Arm/Group | Infliximab 5mg/kg
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab 5mg/kg
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Crohn's Disease Endoscopic Index of Severity (CDEIS) Blinded Score at Week 6
Description: CDEIS endoscopically assesses mucosal status, by summing the following six component scores: number of bowel segments with deep ulcerations divided by number of visualized bowel segments; number of bowel segments with superficial ulcerations divided by number of visualized bowel segments; mean proportion of bowel segment surface involved by disease measured on 0-10 cm visual analog scale (VAS); mean proportion of bowel segment surface area involved by ulcerations measured on 0-10 cm VAS; presence of ulcerated stenosis anywhere; and presence of non-ulcerated stenosis anywhere. An observer who viewed procedural videotape while blinded to the allocation number and visit of the endoscopy scored the CDEIS. The sum of the six components can range from 0-44, with a higher sum indicating greater severity of mucosal inflammation. Change from baseline is defined as Week 6 minus baseline CDEIS scores, with a negative change from baseline indicating improvement.
Time Frame: Baseline and Week 6
Population: Participants who had a blinded CDEIS score at both baseline and at Week 6.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Infliximab 5 mg/kg: Infliximab administered intravenously at a dose of 5 mg/kg at study weeks 0, 2, 6, 14, and 22
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 13
Score on a scale | -4.8 (4.2)

2. Primary Outcome: Change From Baseline in CDEIS Blinded Score at Week 22
Description: CDEIS endoscopically assesses mucosal status, by summing the following six component scores: number of bowel segments with deep ulcerations divided by number of visualized bowel segments; number of bowel segments with superficial ulcerations divided by number of visualized bowel segments; mean proportion of bowel segment surface involved by disease measured on 0-10 cm visual analog scale (VAS); mean proportion of bowel segment surface area involved by ulcerations measured on 0-10 cm VAS; presence of ulcerated stenosis anywhere; and presence of non-ulcerated stenosis anywhere. An observer who viewed procedural videotape while blinded to the allocation number and visit of the endoscopy scored the CDEIS. The sum of the six components can range from 0-44, with a higher sum indicating greater severity of mucosal inflammation. Change from baseline is defined as Week 22 minus baseline CDEIS scores, with a negative change from baseline indicating improvement.
Time Frame: Baseline and Week 22
Population: Participants who had a blinded CDEIS score at both baseline and at Week 22.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 12
Score on a scale | -7.3 (5.5)

3. Primary Outcome: Change From Baseline in Serum High Sensitivity C-reactive Protein (hsCRP) at Week 6
Description: Concentrations of the serum biomarker hsCRP were determined at baseline and at Week 6. The change from baseline was Week 6 minus baseline.
Time Frame: Baseline and Week 6
Population: Participants with measurements for hsCRP at both baseline and at Week 6.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 12
mg/L | -38.1 (30.4)

4. Primary Outcome: Change From Baseline in Serum hsCRP at Week 22
Description: Concentrations of the serum biomarker hsCRP were determined at baseline and at Week 22. The change from baseline was Week 22 minus baseline.
Time Frame: Baseline and Week 22
Population: Participants with measurements for hsCRP at both baseline and at Week 22.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 14
mg/L | -28.0 (39.3)

5. Primary Outcome: Change From Baseline in Stool Calprotectin at Week 6
Description: Concentrations of the stool biomarker calprotectin were determined at baseline and at Week 6. The change from baseline was Week 6 minus baseline.
Time Frame: Baseline and Week 6
Population: Participants with measurements for calprotectin at both baseline and at Week 6.
Measure: Mean (Standard Deviation); unit: µg/g
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 15
µg/g | 231.1 (4099.6)

6. Primary Outcome: Change From Baseline in Stool Calprotectin at Week 22
Description: Concentrations of the stool biomarker calprotectin were determined at baseline and at Week 22. The change from baseline was Week 22 minus baseline.
Time Frame: Baseline and Week 22
Population: Participants with measurements for calprotectin at both baseline and at Week 22.
Measure: Mean (Standard Deviation); unit: µg/g
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 13
µg/g | 98.3 (3236.7)

7. Primary Outcome: Change From Baseline in Serum Lipocalin-2 at Week 6
Description: Concentrations of the serum biomarker lipocalin-2 were determined at baseline and at Week 6. The change from baseline was Week 6 minus baseline.
Time Frame: Baseline and Week 6
Population: Participants with measurements for lipocalin-2 at both baseline and at Week 6.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 15
ng/mL | -103.7 (108.3)

8. Primary Outcome: Change From Baseline in Serum Lipocalin-2 at Week 22
Description: Concentrations of the serum biomarker lipocalin-2 were determined at baseline and at Week 22. The change from baseline was Week 22 minus baseline.
Time Frame: Baseline and Week 22
Population: Participants with measurements for lipocalin-2 at both baseline and at Week 22.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 15
ng/mL | -104.6 (108.9)

9. Primary Outcome: Change From Baseline in Regenerating Islet-Derived 3-Alpha (REG3-A) at Week 6
Description: Concentrations of the serum biomarker REG3-A were determined at baseline and at Week 6. The change from baseline was Week 6 minus baseline.
Time Frame: Baseline and Week 6
Population: Participants with measurements for REG3-A at both baseline and at Week 6.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 14
ng/mL | -20.7 (20.9)

10. Primary Outcome: Change From Baseline in REG3-A at Week 22
Description: Concentrations of the serum biomarker REG3-A were determined at baseline and at Week 22. The change from baseline was Week 22 minus baseline.
Time Frame: Baseline and Week 22
Population: Participants with measurements for REG3-A at both baseline and at Week 22.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 15
ng/mL | -21.2 (30.3)

11. Primary Outcome: Coefficient of Determination (R^2) For Predicting The Change From Baseline In Blinded CDEIS Score From The Changes From Baseline In Four Biomarkers At Weeks 6 and 22
Description: To determine R^2 a multiple linear regression analysis was conducted with the change from baseline in CDEIS score as the response variable and the baseline CDEIS score, changes from baseline in the four biomarkers serum hsCRP, serum lipocalin-2, serum Reg3-A, and stool calprotectin (their concentrations were log-transformed to make the mean function of the response more linear) at Weeks 6 and 22 as the predictor variables. CDEIS scores were provided by a blinded observer who viewed procedural videotape while blinded to the allocation number and visit of the endoscopy. The R^2 can range from 0 to 1; with higher values indicating greater predictability of the model. The primary hypothesis is that the true R^2 at weeks 6 and 22 is approximately 0.7.
Time Frame: Baseline and Week 6 or 22
Population: Participants who had a blinded CDEIS score and measurements for each of the biomarkers included in the models at both baseline and at Week 6 or 22.
Measure: Number; unit: Coefficient of Determination
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 15
Coefficient of Determination
  Week 6 (n = 9) | 0.920 [0.458 to 0.929]
  Week 22 (n = 10) | 0.638 [0.539 to 0.946]
Statistical Analysis 1: Comparison: Infliximab 5 mg/kg; Week 6; Test type: Superiority or Other; p = 0.071, Multiple Linear Regression
Statistical Analysis 2: Comparison: Infliximab 5 mg/kg; Week 22; Test type: Superiority or Other; p = 0.381, Multiple Linear Regression

12. Secondary Outcome: Concordance Correlation Coefficient for Comparison of Repeat Baseline Measurements of Biochemical Biomarkers
Description: Based on two measurements at baseline, the concordance correlation coefficient (CCC) was computed for each of four biomarkers, using a mixed effects model with a fixed factor for repeat measurements and a random factor for participant. The CCC can range from 0 to 1 with higher values indicating greater concordance between the 2 measurements.
Time Frame: Baseline Visit 1 (one week prior to dosing), Baseline Visit 2 (1-2 days prior to dosing)
Population: Participants who had both baseline serum or stool measurements available for analysis.
Measure: Number (90% Confidence Interval); unit: Correlation coefficient
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 15
Correlation coefficient
  serum hsCRP (n=14) | 0.954 [0.913 to 0.995]
  serum REG3-A (n=15) | 0.974 [0.952 to 0.996]
  serum lipocalin-2 (n=15) | 0.910 [0.835 to 0.986]
  stool calprotectin (n=15) | 0.792 [0.629 to 0.954]

13. Secondary Outcome: Concordance Correlation Coefficient for Comparison Between Central Endoscopic Evaluation and Site Endoscopic Evaluation
Description: The CCC of blinded (central) versus unblinded (site) scores from either CDEIS or the Simple Endoscopic Score for Crohn's Disease (SES-CD) was determined at Baseline, Week 6 and Week 22. SES-CD sums the following scores: presence and size of ulcers in five visualized bowel segments; extent of ulcerated surface in five visualized bowel segments; extent of affected surface in five visualized bowel segments; presence and type of narrowings in five visualized bowel segments; and can range from 0-56, with a higher sum indicating greater severity of mucosal inflammation. The CCC can range from 0 to 1 with higher values indicating greater concordance between the 2 measurements.
Time Frame: Baseline, Week 6, Week 22
Population: Participants who had both blinded and unblinded scores available for analysis.
Measure: Number (90% Confidence Interval); unit: Correlation coefficient
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 15
Correlation coefficient
  CDEIS Baseline (n = 15) | 0.662 [0.428 to 0.896]
  CDEIS Week 6 (n = 13) | 0.693 [0.458 to 0.929]
  CDEIS Week 22 (n = 12) | 0.743 [0.539 to 0.946]
  SES-CD Baseline (n = 15) | 0.453 [0.176 to 0.729]
  SES-CD Week 6 (n = 13) | 0.937 [0.879 to 0.995]
  SES-CD Week 22 (n = 13) | 0.753 [0.562 to 0.945]

ADVERSE EVENTS:
Time Frame: From 4 weeks prior to first dose, until 2 weeks after last dose (up to 28 weeks)
Description: All enrolled participants
Groups:
- Pre-study: From 4 weeks prior to first dose, up to first dose of infliximab
- Post-study: From last dose of study drug, up to 24 days after last dose of infliximab
Arm/Group | Pre-study | Infliximab 5mg/kg | Post-study
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/15 | 0/15
Other Adverse Events (participants affected / at risk) | 7/15 | 13/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-study (N=15) | Infliximab 5mg/kg (N=15) | Post-study (N=15)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pre-study (N=15) | Infliximab 5mg/kg (N=15) | Post-study (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0/0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (6) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (7) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, and on the presentation with regard to the following: proprietary information; the accuracy of the information; and that the presentation is fairly balanced and in compliance with FDA regulations.